CLINICAL TRIAL: NCT06778070
Title: National Program to Overcome Pelvic Pain studY (POPPY)
Acronym: POPPY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Stanford University (Other); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-41220; R01AT012461 (NIH)
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pelvic Pain Syndrome (CPPS); Chronic Pelvic Pain Syndrome; Chronic Pelvic Pain
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor yoga program (Experimental): Instruction in the therapeutic yoga intervention will be delivered through 75-minute group classes occurring twice weekly for a 2-month (8-week) intervention instruction period, involving a trained instructor and an expected 6-10 students (a.k.a. participants) using a secure Zoom videoconference platform.
  Following the 8-week intervention instruction period, additional optional once-weekly, 75-minute drop-in group classes will be offered over an additional 8-week intervention maintenance period.
  Interventions: Other: Pelvic floor yoga
- Physical conditioning program (Skeletal muscle stretching and strengthening program) (Active Comparator): The physical conditioning program (skeletal muscle stretching and strengthening program) intervention will begin with a group orientation led by a physical trainer, who will provide an overview of the program. This will be followed by 75-minute twice-weekly group classes, each with an expected class size of 6-10 participants, led by the same physical trainer who has received study-specific training from the study's expert physical therapist consultant, and using a secure Zoom videoconference platform.
  Following the 8-week intervention instruction period, additional optional once-weekly, 75-minute drop-in group classes will be offered over an additional 8-week intervention maintenance period.
  Interventions: Other: Physical conditioning

INTERVENTIONS:
Other: Pelvic floor yoga — Pelvic floor yoga
  Arms: Pelvic floor yoga program
Other: Physical conditioning — Physical conditioning
  Arms: Physical conditioning program (Skeletal muscle stretching and strengthening program)

SUMMARY:
A randomized, parallel-group, investigator-blinded, comparative effectiveness trial of a fully remote, videoconference-based pelvic floor yoga program versus a physical conditioning program for women with chronic pelvic pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Women (individuals reporting female sex assigned at birth who self-identify as women or non-binary) aged 18 years or older
* Report chronic or recurrent pain in the pelvis (between or below the anterior iliac crests) for at least 6 months
* Report at least moderate pain intensity based on a screening pain log
* Report prior clinical evaluation of their pelvic pain by a healthcare professional including at least a superficial pelvic exam
* Willing to refrain from initiating new clinical treatments that may affect their pain during the study period

Exclusion Criteria:

* Report pelvic pain occurring exclusively with menses or exclusively during sexual intercourse (although candidates with at least some pain between menses or intercourse are still eligible)
* Participation in organized yoga classes or muscle strengthening programs (e.g., Pilates) in the past 4 weeks, or any prior yoga therapy specifically directed at pelvic pain
* Lacking technical requirements to complete intervention classes by video, including no access to broadband internet or a Zoom-compatible device larger than a smartphone [display screen at least 7 inches in diagonal] (although the study team may loan devices to participants from underrepresented backgrounds)
* Currently pregnant (by self-report or screening test), pregnant within the past 12 weeks, or planning pregnancy during the study period
* Diagnosed with an alternate, reversible cause of pelvic pain that is unlikely to respond to yoga and requires another treatment modality (e.g., current pelvic infection or a gynecologic dermatosis)
* Surgery or irradiation to the genital or pelvic structures within the past 12 weeks, or anticipating upcoming surgery or irradiation to these structures during the study period
* Initiation, dose escalation, or weaning of pharmacologic agents that may affect pelvic pain severity in the past 4 weeks, such as analgesics, antidepressants, or anticonvulsants-(however, women on stable doses of these medications for at least 4 weeks will still be eligible)
* Use of formal psychological therapies specifically for pelvic pain (e.g., systematic desensitization, cognitive therapy, relaxation therapy) within 4 weeks of screening, or plans to engage in these therapies during the study period
* Unable to walk up a flight of stairs or at least 2 blocks on level ground (i.e., functional capacity < 4 METs), or unable to get up from a supine to a standing position without assistance
* Participation in another interventional study that might interfere with or confound study procedures, or known conflict with multiple upcoming study intervention class dates
* Inability to understand the informed consent form or fill out questionnaires or complete study interviews
* Any other serious physical or mental issue that, in the opinion of the investigators, would interfere with study participation (e.g., advanced dementia, uncontrolled substance use or serious mental illness, life expectancy <6 months)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain intensity "on average" using standard 0-10 numerical rating scale, measured using logs in which participants self-report pain intensity over the past week, and assessed over 4 months of intervention | After 4 months of intervention instruction and maintenance period.
  4 months of intervention (2 months of instruction as well as 2 months of maintenance)
Pelvic pain intensity "at its worst" using standard 0-10 numerical rating scale, measured using logs in which participants to self-report pain intensity over the past week, and assessed over 4 months of intervention | After 4 months of intervention instruction and maintenance period.
  4 months of intervention (2 months of instruction as well as 2 months of maintenance)

SECONDARY OUTCOMES:
Percent of participants achieving reductions in pelvic pain intensity "on average" of at least 30% from baseline (using a standard 0-10 numerical rating scale) after 4 months of intervention | After 4 months of intervention instruction and maintenance period.
  4 months of intervention (2 months of instruction as well as 2 months of maintenance)
Percent of participants achieving reductions in pelvic pain intensity "at its worst" of at least 30% from baseline (using a standard 0-10 numerical rating scale) after 4 months of intervention | After 4 months of intervention instruction and maintenance period.
  4 months of intervention (2 months of instruction as well as 2 months of maintenance)
Psychological impact of chronic pelvic pain, measured by the psychological domain score of the Impact of Female Chronic Pelvic Pain Questionnaire (IF-CPPQ) over 4 months of intervention | After 4 months of intervention instruction and maintenance period.
  4 months of intervention (2 months of instruction as well as 2 months of maintenance)
Sexual impact of chronic pelvic pain, measured by the sexual domain score of the Impact of Female Chronic Pelvic Pain Questionnaire (IF-CPPQ) over 4 months of intervention | After 4 months of intervention instruction and maintenance period.
  4 months of intervention (2 months of instruction as well as 2 months of maintenance)
General interference of pain with daily functioning in women with CPPS, as measured by scores on the PROMIS Pain Interference 4a measure from baseline to 4 months of intervention | After 4 months of intervention instruction and maintenance period.
  4 months of intervention (2 months of instruction as well as 2 months of maintenance.
Perceived stress as measured by scores on the 4-item Perceived Stress Scale over the 4-month intervention period | After 4 months of intervention instruction and maintenance period.
  4-month intervention period (2 months of intervention instruction and 2 months of maintenance)
Sleep quality as measured by scores on the PROMIS Sleep Disturbance Short Form over the 4-month intervention period | After 4 months of intervention instruction and maintenance period.
  4-month intervention period (2 months of intervention instruction and 2 months of maintenance).
Pelvic problems-related sexual function as measured by scores on the Pelvic Problems Interference subscale of the Sexual Health Outcomes in Women Questionnaire (SHOW-Q) over the 4-month intervention period | After 4 months of intervention instruction and maintenance period.
  4-month intervention period (2 months of intervention instruction and 2 months of maintenance)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, Principal Investigator — University of California, San Francisco; Carolyn Gibson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes